CLINICAL TRIAL: NCT07170358
Title: Screening of Diagnostic Biomarkers and Related Mechanisms for Radiation-induced Xerostomia
Brief Title: Screening of Biomarkers and Related Mechanisms for RIX
Acronym: RIX
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: The Tumor Hospital of Jiangsu Province (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Jinling Hospital Affiliated to Nanjing University School of Medicine (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2025-0461
Record Dates: First submitted 2025-09-07; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-07

CONDITIONS: Xerostomia Due to Radiotherapy (Disorder)
Keywords: Head and neck tumor; radiotherapy; biomarkers; xerostomia
MeSH Terms: conditions — Head and Neck Neoplasms; Xerostomia | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — Serum, plasma, blood cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- No xerostomia before radiotherapy: Resting saliva flow rate greater than 1ml/10min before radiotherapy
- Mild xerostomia during radiotherapy: During radiotherapy, a resting saliva flow rate between 0.5ml/10min-1ml/10min is considered mild dry mouth
  Interventions: Radiation: Radiation Therapy
- Moderate to severe xerostomia during radiotherapy: A resting saliva flow rate below 0.5ml/10min during radiotherapy is considered moderate to severe xerostomia
  Interventions: Radiation: Radiation Therapy
- Mild xerostomia after radiotherapy: After radiotherapy, a resting saliva flow rate between 0.5ml/10min-1ml/10min is considered mild dry mouth
  Interventions: Radiation: Radiation Therapy
- Moderate to severe xerostomia xerostomia after radiotherapy: A resting saliva flow rate below 0.5ml/10min after radiotherapy is considered moderate to severe xerostomia
  Interventions: Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Radiation Therapy — Radiotherapy for Head and Neck Cancer Patients
  Groups: Mild xerostomia after radiotherapy; Mild xerostomia during radiotherapy; Moderate to severe xerostomia during radiotherapy; Moderate to severe xerostomia xerostomia after radiotherapy

SUMMARY:
A large number of patients undergoing radiotherapy and chemotherapy are suffering from dry mouth. Due to reduced saliva secretion, patients may experience symptoms such as difficulty chewing and swallowing. In severe cases, they may also experience pain and burning sensation in the oral mucosa, decreased taste, ulcers, which seriously affect the quality of life of patients. However, radiation-induced dry mouth lacks early objective predictive indicators (molecular biomarkers) and the mechanism is unclear. Only when patients experience clinical symptoms will symptomatic treatment be taken to alleviate them. Therefore, elucidating the mechanism of radiation-induced dry mouth syndrome (RIX) and achieving early prediction, detection, and intervention of RIX are crucial in improving the prognosis and quality of life of radiotherapy patients. It is urgent to seek early and precise detection targets in clinical practice to predict dry mouth caused by irreversible damage to salivary gland tissue. This study aims to collect blood samples from patients with severe dry mouth before and after radiotherapy and chemotherapy in clinical practice. Multiple omics techniques will be used to search for predictive molecular biomarkers for RIX, construct a predictive model, and verify the sensitivity and specificity of the biomarkers. The goal is to predict the occurrence of RIX early in clinical practice, intervene in advance, greatly improve the prognosis of radiotherapy and chemotherapy patients, and enhance their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of head and neck cancer;
* Plan to undergo curative treatment with radiotherapy alone or in combination with synchronous chemotherapy, immunotherapy, or targeted therapy;
* Age greater than or equal to 18 years old, Fully understand the purpose and significance of this study, voluntarily participate and sign an informed consent form.

Exclusion Criteria:

* Metastatic diseases;
* History of head and neck radiotherapy;
* Severe dry mouth before radiotherapy;
* Suffering from advanced chronic diseases: heart failure - New York Heart Association functional classification III/IV, renal failure - estimated glomerular filtration rate under 30mL/min/1.73m2, liver failure - Child Pugh score C or D.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Head and neck cancer radiotherapy patients
Sampling Method: Non-Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2024-05-17 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Resting saliva flow measurement | From the start of radiotherapy to 3 months after completion
  When fasting in the morning, instruct the patient to gather saliva at the bottom of the mouth, lower their head and slightly open their mouth to allow the gathered saliva to naturally flow into the oral cup. Generally, collect for 10 minutes, with less than 1ml indicating mild dry mouth, less than 0.5ml indicating moderate dry mouth, and less than 0.1ml indicating severe dry mouth.

SECONDARY OUTCOMES:
Changes in Quality of Life and xerostomia Questionnaire Scores | From the start of radiotherapy to 3 months after completion
  According to the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-head and neck35(EORTC QLQ-H&N35) questionnaire, dry mouth symptoms were scored and classified in patients with postoperative oral dryness after radiotherapy.In the dry mouth category, responses of "quite a bit" and "very much" and a total score difference of ≥ 10 points before and after treatment are defined as moderate to severe dry mouth.The higher the overall score, the worse the situation.
Comparison of Body Mass Index | From the start of radiotherapy to 3 months after completion
  Measure the weight changes of patients before and after radiotherapy, weight and height will be combined to report BMI in kg/m^2.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Affiliated Jinling Hospital, Medical School of Nanjing University, Nanjing, Jiangsu
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No